CLINICAL TRIAL: NCT05890326
Title: Pain Neuroscience Education and Motor Imagery-based Exercise Protocol in Fibromyalgia
Brief Title: Pain Neuroscience Education and Motor Imagery-based Exercise Protocol for Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Mesut Karahan, Assoc. Prof., Uskudar University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: fibromyalgiaUSK
Record Dates: First submitted 2023-05-16; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Fibromyalgia; Pain; Psychology Regression
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): No intervention was applied to fibromyalgia patients in this group. This was because it was a control group that would evaluate the effects on outcomes by comparing them with other intervention (behavioral) groups.
- Motor imagery-based exercise protocol (MIEP) (Experimental): Motor imagery-based exercise protocol (MIEP) applied in this group.
  Interventions: Behavioral: Motor imagery-based exercise protocol (MIEP)
- Pain neuroscience education (PNE) (Experimental): Pain neuroscience education (PNE) applied in this group.
  Interventions: Behavioral: Pain neuroscience education (PNE)
- Combination Group (Active Comparator): Both Pain neuroscience education (PNE) and Motor imagery-based exercise protocol (MIEP) applied in this group.
  Interventions: Behavioral: Combination Group

INTERVENTIONS:
Behavioral: Pain neuroscience education (PNE) — Pain neuroscience education (PNE) is a health education intervention that aims to provide up-to-date information on neuroscience developments in the field of chronic pain. All patients were trained once a week for 12 weeks, in groups of 3-4 people, for a maximum of 6 sessions and a minimum of 60 minutes. During the intervention, psychological factors such as self-efficacy, pain intervention/injury, coping with pain, catastrophic thoughts, emotional response to pain, anxiety, frustration/anger, fear of harm, concerns about pain, and fear of pain were examined. and discussed with patients. The sessions aimed to provide patients with a better understanding of their chronic pain by addressing the multifactorial aspects of chronic pain, sensitization and the plasticity of the brain, thus involving patients in treatment.
  Arms: Pain neuroscience education (PNE)
Behavioral: Motor imagery-based exercise protocol (MIEP) — All patients performed sessions of maximum 60 minutes in groups of 3-4 people twice a week for 12 weeks. This study protocol was developed in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. The key standard was to practice simple and safe exercises that would encourage the patient to repeat the program at home. The exercises proposed in MIEP were selected according to the following principles: slowness, painlessness, arousing attention, easy to imagine. The main purpose of the motor imagery exercises was to bring the patient back to the state of "feeling and self-perception" of the execution of the movement. More important than the "quantity" of repetition was the painless "quality" of movement. It was performed in 3 phases: relaxation (3 minutes), MI (8.5 minutes per image) and refocus (3 minutes), which included both kinesthetic imagery (KI) and visual imagery (VI).
  Arms: Motor imagery-based exercise protocol (MIEP)
Behavioral: Combination Group — Subjects received 6 sessions of Pain neuroscience education (PNE) and 12 weeks (2 times a week) of Motor imagery-based exercise protocol (MIEP).
  Arms: Combination Group

SUMMARY:
The main aim of this study is to find out whether applying both pain neuroscience education (PNE) and motor imagery-based exercise protocol (MIEP) will primarily reduce the pain of fibromyalgia. These therapies could show an evidence of improvement in fibromyalgia patients. However, there are no studies evaluating their effectiveness in combination.

Secondary outcomes:

To assess motor imagery ability of PNE in fibromyalgia patients

To assess motor imagery ability of MIEP in fibromyalgia patients

To evaluate the motor imagery ability of PNE+MIEP combined in fibromyalgia patients

To evaluate pain beliefs of PNE in fibromyalgia patients

To assess the pain beliefs of MIEP in fibromyalgia patients

Combined PNE+MIEP to assess pain beliefs in fibromyalgia patients.

To assess fear of movement in fibromyalgia patients of PNE

To assess fear of movement in fibromyalgia patients of MIEP

Combined PNE+MIEP to assess fear of movement in patients with fibromyalgia

PNE to assess anxiety, depression, cognitive and mood in patients with fibromyalgia.

To assess anxiety, depression, cognitive and mood in patients with fibromyalgia MIEP

To evaluate anxiety, depression, cognitive and mood in patients with fibromyalgia together with PNE+MIEP

PNE to assess self-esteem and body awareness in fibromyalgia patients.

To assess self-esteem and body awareness in fibromyalgia patients of MIEP

Combined PNE+MIEP to assess self-esteem and body awareness in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing widespread chronic pain for more than 12 months
* Pain in at least 12 or more of 18 tender points with a pressure of 5 kg/cm2
* 18 to 60 years old
* Not using pharmacological therapeutics
* Not having participated in any pain program.
* Not having participated in any physical exercise programs in the last twelve

Exclusion Criteria:

* Pregnancy
* Not being able to do a physical activity program
* Currently receiving treatment with any alternative medical methods (eg.hyperbaric).
* Cardiovascular, psychiatric, autoimmune, cancer, etc. children with secondary different disease
* Other causes of chronic pain
* Receiving any treatment support related to pain
* Mental disability status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 12 weeks
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  HADS - One questionnaire, comprising of fourteen questions The questionnaire features seven questions for anxiety and seven for depression of which can be answered within 2 - 5 minutes. Responses are scored on a scale of 3 to 0 - The maximum score is therefore 21 for Anxiety and 21 for Depression.
  Odd numbers: 1, 3, 5, 7, 9, 11 and 13 are Anxiety Questions (Grey in Colour) Even numbers: 2, 4, 6, 8, 10, 12 and 14 are Depression Questions (White in Colour)
  The two sub-scales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into four stages:
  Scores of: 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
The Motion Imagery Questionnaire-3 (HLFS-3) | 12 weeks
  The Motion Imagery Questionnaire-3 (HLFS-3) is an adaptation of the Motion Imagery Questionnaire. It consists of 3 subscales and a total of 12 items evaluating external visual imagery, internal visual imagery and kinesthetic imagery. Before starting the evaluation, the participants were given the necessary information about the survey. Each of the 12 tasks in the questionnaire was first performed physically, then the participant returned to the starting position and imaged according to the desired imagery type.
  Scoring was made between 1 and 7, with 1 point: very difficult to see/feel, 7 points: very easy to see/feel. While calculating the score, the internal visual imagery, external visual imagery and kinesthetic imagery scores were added separately and averaged by dividing by 4. As a result, the score of each subscale was obtained.
The Pain Beliefs Questionnaire (PBQ) | 12 weeks
  The Pain Beliefs Questionnaire (PBQ), a 32-item self-report measure of the pain beliefs of children and adolescents with chronic pain, assesses cognitive appraisals that may influence children's coping strategies, disability, mood, and pain severity. For each item on the PBQ, respondents indicate how true the statement is on a 5-point rating scale ranging from "not at all true" (0) to "very true" (4). Subscale total scores are computed by averaging items pertaining to each subscale.
The Pain Catastrophizing Scale (PCS) | 12 weeks
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain. Patients are asked to rate the degree to which they have any of the thoughts described in the questionnaire using a 5-point Likert scale ranging from 0 (never) to 4 (always). The total score is the sum of the scores for the individual items, and ranges from 0 to 52.
The Tampa Scale for Kinesiophobia (TSK) | 12 weeks
  The Tampa Scale for Kinesiophobia (TSK) is a 17-item questionnaire that quantifies fear of movement. Individual item scores range from 1-4, with the negatively worded items (4,8,12,16) having a reverse scoring (4-1). The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Adapting the Scale of Cognitive Emotion Regulation Strategies | 12 weeks
  The scale aims to determine the level of cognitive emotion regulation strategies used by a person against a particular event or events in general, regardless of clinical or non-clinical distinction. The scale, consisting of 36 items and 9 sub-dimensions, has a five-point Likert-type rating (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always). There are 4 items in each sub-dimension and the lowest score from a sub-dimension is 4 and the highest score is 20.
Rosenberg Self-esteem Scale | 12 weeks
  Rosenberg self-esteem scale is: The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.
The Body Awareness Questionnaire | 12 weeks
  The body awareness questionnaire is a 18 item scale, with the total scale score calculated as a sum of the items. Items are scored on a 1-7 scale, with the total scale score calculated as a sum of the items. The questions with asterisks are reverse scored.

CONTACTS AND LOCATIONS:
Overall Officials: Selin Kırcali, Msc, Study Director — Üsküdar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)